CLINICAL TRIAL: NCT06453746
Title: Effectiveness of Dementia Prevention in Elderly Patients With Mild Cognitive Impairment at Nhân dân Gia Định Hospital, Hồ Chí Minh City
Brief Title: Effectiveness of Non-pharmacological Interventions for Dementia Prevention in Elderly Patients With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 625/HĐĐĐ-ĐHYD
Record Dates: First submitted 2024-05-31; First posted 2024-06-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mild Cognitive Impairment; Dementia Prevention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based cognitive training exercises (Active Comparator): The cognitive training exercises program includes a total of 19 exercises and activities. The 19 exercises are divided into 8 groups: (1) warm up and cool down (relaxation exercise), (2) episodic memory, (3) digit span and calculation, (4) language, (5) Linking Letters & Numbers, (6) Imagery, (7) Visuoconstructional skills, (8) linking ADL/IADL tasks.
  Subjects are provided with 19 exercises and instructed to perform them at home. Home-based exercises will be assessed weekly. Subjects are provided with a logbook to track their progress with the home exercises and were given the opportunity to provide feedback, ask questions, and receive support for any difficulties encountered during the process.
  All cognitive training exercises are based on the Technical Procedure Instructions issued by the Vietnamese Ministry of Health.
  Interventions: Other: Home-based cognitive training exercises
- Supervised cognitive training exercises (Experimental): The cognitive training exercises program includes a total of 19 exercises and activities. The 19 exercises are divided into 8 groups: (1) warm up and cool down (relaxation exercise), (2) episodic memory, (3) digit span and calculation, (4) language, (5) Linking Letters & Numbers, (6) Imagery, (7) Visuoconstructional skills, (8) linking ADL/IADL tasks.
  The subjects are given exercises at the hospital under the supervision of physiotherpist/ physiatrist, and are also instructed to do the exercises at home.
  Home-based exercises will be assessed weekly. Subjects are provided with a logbook to track their progress with the home exercises and were given the opportunity to provide feedback, ask questions, and receive support for any difficulties encountered during the process.
  All cognitive training exercises are based on the Technical Procedure Instructions issued by the Vietnamese Ministry of Health.
  Interventions: Other: Supervised cognitive training exercises

INTERVENTIONS:
Other: Home-based cognitive training exercises — The subjects received (i) education on lifestyle modification, (ii) home-based cognitive training exercises with physiotherapist/ physiatrist contact when needed and (iii) a physical training exercises conducted at hospital under the supervision of physiotherapist/ physiatrist (3 weekly session for 12 weeks).
  This arm has a duration of 12 weeks.
  Arms: Home-based cognitive training exercises
Other: Supervised cognitive training exercises — The subjects received (i) education on lifestyle modification, (ii) supervised cognitive training exercises at hospital (1 weekly session for 12 weeks) and (iii) a physical training exercises conducted in a hospital under the supervision of physiotherapist/ physiatrist (3 weekly session for 12 weeks).
  This arm has a duration of 12 weeks.
  Arms: Supervised cognitive training exercises

SUMMARY:
The aims of this study is to evaluate the effectiveness of non-pharmacological interventions program in preventing progression from mild cognitive impairment to dementia in patients with mild cognitive impairment in the short term, at Nhân dân Gia Định Hospital, Hồ Chí Minh City.

DETAILED DESCRIPTION:
A non-pharmacological interventions program in dementia prevention is highly promising because: (i) the results of using drugs (e.g. cholinesterase inhibitors) have not been successful, so non-pharmacological interventions may be a promising and risk-free alternative; (ii) people with mild cognitive impairment still maintain memory capacity that allows them to learn and apply new information and skills; (iii) interventions at an early stage of the cognitive decline process will bring maximum benefits; (iv) there is evidence that cognitive training exercises have a positive effect on cognitive decline and are one of protective factors against dementia.

Although studies on non-pharmacological prevention programs with cognitive training exercises as a key component are not uncommon, we found that there are still some unclear points. First and foremost, there has been no cognitive training exercises in Vietnamese that has been studied. Most use foreign language communication, making language-related stimuli inapplicable in Vietnam. Next, the exercise design either focuses on improving thinking and flexibility, which is more suitable for younger people, or only prioritizes impacting certain cognitive domains. Finally, many current programs are integrated as technology applications on phones, which, although convenient, are not really user-friendly for the elderly in Vietnam due to habits, operating system response delays, and equipment costs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with mild cognitive impairment:

  * Cognitive complaints from the subject or a family member.
  * Report a decline in cognitive function compared to the subject's previous ability over the past year OR
  * Evidence from clinical assessment, specifically here is MMSE screening with results of 24-29 points.
  * Subjects did not suffer major impacts from cognitive complaints on daily life.
  * No prior diagnosis of dementia.
* Ensure transportation from living location to hospital.
* Have at least one relative or caregiver who can supervise the subject's daily activities.
* Stable chronic underlying conditions (diabetes, hypertension).
* Consent to participate in the study.

Exclusion Criteria:

* Don't know Vietnamese writing.
* Audio-visual ability does not meet the requirements of assessment tests and prevention programs.
* Systemic diseases are contraindications/ restriction to participation in programs and/or cause secondary cognitive impairment (traumatic brain injury, stroke, brain tumor, parkinsonism, epilepsy, acute coronary artery disease, acute myocardial infarction, bone fractures...).
* The assessment score on the Geriatric Depression Scale (GDS-15) is ≥ 5 points.
* Diagnosed with other mental disorders that may limit the ability to understand, communicate and work in groups (schizophrenia, mania, bipolar disorder, dissociative disorder, generalized anxiety disorder).
* Currently participating in another research program on dementia prevention or a research program on medication to prevent dementia within the last 3 months.
* Taking medications that may affect cognitive function, such as benzodiazepines, hypnotics, and antipsychotics.
* Alcohol abuse: drinking alcohol daily or consuming more than 14 units of alcohol per week (equivalent to 10 grams of ethanol, as defined by the Ministry of Health); diagnosed with alcohol dependence or currently being treated for mental illness due to alcohol dependence.
* Do not agree to participate in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Intervention Program | Measured at month 3 and 6 after randomisation
  Evaluating the effectiveness of preventing progression from mild cognitive impairment to dementia using the Montreal Cognitive Assessment (The MoCA Test) in patients with mild cognitive impairment in the short term. Higher scores mean a better outcome. The following result ranges may indicate cognitive impairment: 18-25 points: Mild cognitive impairment. 10-17 points: Moderate cognitive impairment. Fewer than 10 points: Severe cognitive impairment.

SECONDARY OUTCOMES:
Change in Activities of Daily Living | Baseline, Week12, Week24
  Evaluating improvement using The Lawton Instrumental Activities of Daily Living Scale (IADL). Higher scores mean a better outcome.
Change in physical fitness | Baseline, Week12, Week24
  Evaluating improvement using The Senior Fitness Test Kit (Chair stand test, Arm curl test, Step in place test, Up and go test). Higher scores mean a better outcome (except Up and go test).
Change in mental health | Baseline, Week12, Week24
  Evaluating improvement using Geriatric Depression Scale-15 (GDS15). Higher scores mean a worse outcome.
Patient Adherance | Week12
  Adherence is assessed considering the number of individuals who have accepted to participate in the study relative to the number of participants who are recruited. Low < 80%, moderate 80-90%, high > 90%
Patient Attendance | Week12
  Attendance rate is calculated as a percentage of the number of exercise sessions completed by participants by the full amount of sessions they are expected to perform throughout the study. Not achieved < 90%

CONTACTS AND LOCATIONS:
Locations (1):
- Nhân dân Gia Định Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in dementia prevention. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).